CLINICAL TRIAL: NCT07248280
Title: Adding Aprepitant to a Multimodal Strategy for the Prevention of Postoperative Nausea and Vomiting in High-risk Outpatient Surgical Patients
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2026-13145
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Nausea and Vomiting, Postoperative; Prevention
Keywords: Ambulatory care; Aprepitant
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Aprepitant

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, phase III superiority clinical trial conducted in parallel groups with triple blinding
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aprepitant (Experimental): Participants will receive a 40 mg capsule of aprepitant, in addition to standard antiemetic prophylaxis.
  Interventions: Drug: Aprepitant 40mg
- Placebo (Placebo Comparator): Participants will receive a 40 mg capsule of placebo, in addition to standard antiemetic prophylaxis
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aprepitant 40mg — Just before the patient is taken to the operating room, a single oral capsule of 40 mg of aprepitant will be given to the participant to evaluate the effectiveness of 40 mg of aprepitant in preventing postoperative nausea and vomiting (PONV) in outpatient surgery. The protocol was chosen to determine whether adding aprepitant to a standard multimodal strategy provides a clinically measurable benefit compared to placebo.
  Arms: Aprepitant
Drug: Placebo — Just before the patient is taken to the operating room, a single oral capsule of 40 mg of placebo will be given to the participant.
  Arms: Placebo

SUMMARY:
Postoperative nausea and vomiting (PONV) are a frequent and debilitating complications after surgery, affecting up to 80% of patients at high risk in the absence of prophylaxis.

Despite the rigorous application of the recommendations from the American Society of Anesthesiologists (ASA) at CHUM, a recent local study reveals a prevalence of 25% PONV at home after outpatient surgery. However, the therapeutic options at home remain limited.

This study aims to evaluate if the addition of 40 mg aprepitant to a multimodal strategy for preventing PONV improves clinical outcomes in high-risk patients undergoing outpatient surgery.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) are common and debilitating complications that can occur after surgery. Their incidence is estimated to be around 30% in the general population and may reach up to 80% in high-risk patients in the absence of prevention, thus constituting a frequent and major source of dissatisfaction. In outpatient surgery, it is still assumed that postoperative outcomes are straightforward. However, this perception is based on a bias of ignorance, as postoperative outcomes are rarely measured after hospital discharge. However, recent studies suggest that nearly 40% of patients may present with PONV once at home. The symptoms are sometimes considered more debilitating than the postoperative pain itself. Although rarely serious, they have a considerable impact on patient satisfaction and the length of their recovery. In some studies, they even represent the main cause of readmission after outpatient surgery or failure of discharge, resulting in additional costs for the healthcare system.

This study aims to evaluate if the addition of 40 mg aprepitant to a multimodal strategy for preventing post operative nausea and vomitting improves clinical outcomes in high-risk patients undergoing outpatient surgery.

The primary objective of this study is to evaluate the complete response rate, defined as the absence of nausea, vomiting, or the need for rescue treatment within 48 hours following surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over, requiring an ambulatory surgery
* at high risk of post-operative nausea and vomitting defined by at least 3 factors from the Apfel score, calculated just prior to the surgery (female sex; non smoker; previous nausea or vomitting post-op., or motion sickness; expected opioid consumption in postoperative care).

Exclusion Criteria:

* Refusal or unable to consent
* Suspected or documented allergy to aprepitant (emend)
* Concomitant use of medication interacting via the cytochrome CYP3A4 with aprepitant (pimozide, terfenadine, astemizole, comtadin or cisapride).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2026-02-24 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Rate of complete response according to postoperative nausea and vomitting | 48 hours after the surgery
  The rate of 'complete response' (CR), defined as the proportion of patients who experienced no episodes of postoperative nausea or vomiting (PONV) and did not require rescue medication following the addition of 40mg of aprepitant to a multimodal prevention strategy for PONV in high-risk patients during the first 48 hours following surgery.

SECONDARY OUTCOMES:
Severity and frequence of nausea and vomiting | At discharge from recovery room, usually 1h after the end of the surgery, 24 hours and 48 hours after the surgery
  The severity of nausea will be assessed using a questionnaire called the Simplified Postoperative Nausea and Vomitting Severity Score (SPONVSS) which indicates the number of episodes of vomiting and regurgitations from 0 to 4, where 0 represents none, 1, 2 and 3 are the number of episodes and 4 being 4 episodes or more, at three different time points (upon discharge from the recovery room, at 24 and 48 hours after surgery).
Medical economic impact | 48 hours after the surgery
  The medical economic impact will be evaluated in terms of cost-effectiveness by analyzing the hospital admission conversions from ambulatory to inpatient admission, calls to 811 for health advice or the CHUM Patient Health Line, returns to the emergency room, and unplanned medical consultations for reasons exclusively related to PONV. A Willingness to pay questionnaire with one hypothetical question will also be asked 48 hours after surgery.
Quality of recovery | Change between baseline (before surgery) and 48 hours after the surgery
  QoR15 is a valid questionnaire to measure the quality of recovery after surgery and anaesthesia, which includes 15 questions. Each of the 15 items are scored by the patient from 0 (worst score) to 10 (optimal score), giving a lowest possible score of 0 (worst outcome), and a highest possible score of 150 (optimal outcome).
Incidence of side effects | 48 hours after the surgery
  The potential side effects related to the medication, such as fatigue, dizziness, headaches, abdominal bloating, dyspepsia, hiccups, constipation, or diarrhea will be collected.
Patient satisfaction | 48 hours after the surgery
  The overall patient satisfaction will be assessed on a visual analog scale from 0 to 10, where 0 represents completally unsatisfied and 10 represents fully satisfied.
Analgesic consumptions (Opioid and non opioid) | 48 hours after the surgery
  The total opioid consumption will be recorded and expressed in morphine equivalent dose and the consumption of acetaminophen and nonsteroidal anti-inflammatory drugs will also be documented

CONTACTS AND LOCATIONS:
Overall Officials: Maxim Roy, MD, FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No